CLINICAL TRIAL: NCT07044271
Title: An Open-Label, Randomized, 3-Way Crossover Study Comparing the Pharmacokinetics of Multiple Olomorasib (LY3537982) Capsules
Brief Title: A Study of Multiple Olomorasib (LY3537982) Capsules in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 27282; J3M-OX-JZQK (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-06-26; First posted 2025-06-29 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: 3-way crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Olomorasib - (Test Formulation 1) (Experimental): Olomorasib administered orally
  Interventions: Drug: Olomorasib
- Olomorasib - (Test Formulation 2) (Experimental): Olomorasib administered orally
  Interventions: Drug: Olomorasib
- Olomorasib - (Reference Formulation) (Active Comparator): Olomorasib administered orally
  Interventions: Drug: Olomorasib

INTERVENTIONS:
Drug: Olomorasib — Single dose
  Other Names: LY3537982

SUMMARY:
The main purpose of this study is to measure how much olomorasib gets into the bloodstream and how long it takes the body to get rid of it. Healthy participants will take olomorasib by mouth. The study will last about 7 weeks and will include 10 back-to-back overnight stays in the research center.

ELIGIBILITY:
Inclusion Criteria:

* Healthy status as defined by the absence of evidence of any clinically significant active or chronic disease
* Body mass index (BMI): 18.0 to 30.0 kilograms per square meter (kg/m²), inclusive
* Participants assigned male at birth (AMAB) or assigned female at birth (AFAB) who are individuals not of childbearing potential (INOCBP).

Exclusion Criteria:

* Females who are lactating or of childbearing potential
* Clinically significant history of any drug sensitivity, drug allergy, or food allergy
* Have used or plan to use medication within 14 days or 5 half-lives, whichever is longest, prior to admission, with the exception occasional acetaminophen at doses less than or equal to 2 g/day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration versus Time Curve from Time Zero to Time t (AUC[0-tlast]) of Olomorasib | From Day 1, Predose up to 72 hours Postdose
  PK: AUC(0-tlast) of Olomorasib
PK: Area Under the Concentration versus Time Curve from Zero to Infinity (AUC[0-∞]) of Olomorasib | From Day 1, Predose up to 72 hours Postdose
  PK: AUC(0-∞) of Olomorasib
PK: Maximum Observed Drug Concentration (Cmax) of Olomorasib | From Day 1, Predose up to 72 hours Postdose
  PK: Cmax of Olomorasib

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - ICON Early Phase Services, San Antonio, Texas
  - ICON, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No